CLINICAL TRIAL: NCT00419380
Title: Treatment of Clogged Tympanostomy Tubes: An Off-Label Use of Dornase Alfa (Pulmozyme®)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 06-0556; BB-IND Number: 100242
Record Dates: First submitted 2007-01-04; First posted 2007-01-08 (Estimated); Results first posted 2015-03-27 (Estimated); Last update posted 2015-03-27 (Estimated); Status verified 2015-03

CONDITIONS: Otitis Media
Keywords: clogged ear tubes
MeSH Terms: conditions — Otitis Media | interventions — dornase alfa

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- dornase alfa (Pulmozyme®) (Active Comparator): dornase alfa - Pulmozyme®: 5 drops twice daily for 7 days to the affected ear.
  Interventions: Drug: dornase alfa (Pulmozyme®)
- Ofloxin (Active Comparator): Ofloxin : 5 drops twice daily for 7 days to the affected ear.
  Interventions: Drug: dornase alfa (Pulmozyme®)

INTERVENTIONS:
Drug: dornase alfa (Pulmozyme®) — This study will compare two treatment arms. Patients will be randomized to either traditional treatment (Ofloxin)or to experimental treatment [dornase alfa (Pulmozyme®)]. Each arm will have subjects instilling 5 drops twice daily for 7 days to the affected ear.

SUMMARY:
The purpose of this study is to evaluate Pulmozyme® (dornase) as compared to a standard ear drop Floxin® (ofloxicin) to dissolve clogged tubes. This study will monitor the use of the new drug for any problems related to the medication. Patients are being asked to be in this study because they had tubes placed for the treatment of chronic ear infection and the tube(s) are now clogged. Clogged tubes are a common problem found in children with tubes. This problem occasionally is improved with ear drops like Floxin®. However, it is frequently not improved even after this standard ear drop treatment.

DETAILED DESCRIPTION:
The success in treating blocked tubes may relate to the ability to dissolve the material clogging the tube as well as dealing with the thick fluid in the middle-ear. The reasoning behind this study is that the use of Pulmozyme® may be able to treat both of these problems. Pulmozyme® was approved by the FDA in 1994 for the treatment of cystic fibrosis patients. Infections present in airway (lung) secretions of cystic fibrosis patients and the material that plugs ear tubes are in some ways the same. "Off-label" use of a drug is the practice by physicians to use a FDA-approved drug in treating conditions other than what the original approval was intended for. Pulmozyme® has been used to treat other lung diseases not related to cystic fibrosis. There has been no published report on the use of Pulmozyme® to treat ear infections. This study is a clinical trial that compares two treatments and will last for 3 months.

ELIGIBILITY:
Inclusion Criteria:

* subjects from age 1 to 18 years who have undergone tube placement in the previous 9 months.
* subjects with middle-ear fluid on entry into the study will be required to have had a prior normal hearing test.

Exclusion Criteria:

* subjects with symptoms of an acute otitis media (otalgia or otorrhea), sensorineural hearing loss,cranio-facial syndromes, cystic fibrosis, prior ear surgery except tube placement, sensitivity to fluoroquinolones and presence of granulation tissue in the lumen of the tympanostomy tubes will be excluded.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2007-01; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenny H Chan, MD, Principal Investigator — The Children's Hospital
Locations (1):
- The Children's Hospital, Denver, Colorado, United States

REFERENCES:
- [Derived] Chan KH, Allen GC, Kelley PE, Streubel SO, Friedman NR, Yoon P, Gao D, Ruiz AG, Jung TTK. Dornase Alfa Ototoxic Effects in Animals and Efficacy in the Treatment of Clogged Tympanostomy Tubes in Children: A Preclinical Study and a Randomized Clinical Trial. JAMA Otolaryngol Head Neck Surg. 2018 Sep 1;144(9):776-780. doi: 10.1001/jamaoto.2018.1101. PMID 30073253

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dornase Alfa (Pulmozyme®) | Ofloxin
Started | 19 | 22
Completed | 18 | 12
Not Completed | 1 | 10
Not completed — Lack of Efficacy | 1 | 7
Not completed — Physician Decision | 0 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dornase Alfa (Pulmozyme®) | Ofloxin | Total
Number analyzed (Participants) | 19 | 22 | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 19 | 22 | 41
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 4.45 (3.30) | 4.05 (2.27) | 4.24 (2.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 10
  Male | 13 | 18 | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 1 | 5
  Not Hispanic or Latino | 15 | 21 | 36
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 19 | 20 | 39
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 19 | 22 | 41

OUTCOME MEASURES:

1. Primary Outcome: Patency of the Tympanostomy Tube at the Day-14 Visit.
Time Frame: 14 days
Population: Analysis performed on ear level. Some participants received drops in both ears and thus both ears were included in analysis.
Measure: Number; unit: Ear
Groups:
- Dornase Alfa (Pulmozyme®): dornase alfa (Pulmozyme®): 5 drops twice daily for 7 days to the affected ear. Right ear n=8; Left ear n= 15
- Ofloxin: Ofloxin: 5 drops twice daily for 7 days to the affected ear. Right ear n=11; Left ear n=12
Arm/Group | Dornase Alfa (Pulmozyme®) | Ofloxin
Number analyzed (Participants) | 19 | 18
Ear
  Right Ear | 8 | 11
  Left Ear | 15 | 12
Statistical Analysis 1: Comparison: Dornase Alfa (Pulmozyme®) vs Ofloxin; Two by two contingency table was used to compare our outcome, tube patency yes/no, by our two independent variables, dornase alfa (Pulmozyme®) and Ofloxin; Test type: Superiority or Other; p = .36, Chi-squared

2. Secondary Outcome: Presence or Absence of Drainage in the Ear Canal and Fluid in the Middle Ear at the the Day-14 Visit.
Description: Outcome measure data table represents the absence of drainage at day- 14
Time Frame: 14 days
Measure: Number; unit: Ear
Arm/Group | Dornase Alfa (Pulmozyme®) | Ofloxin
Number analyzed (Participants) | 19 | 18
Ear
  Right Ear | 8 | 11
  Left Ear | 15 | 12
Statistical Analysis 1: Comparison: Dornase Alfa (Pulmozyme®) vs Ofloxin; Test type: Superiority or Other; p = .26, Chi-squared — Two by two contingency table was used to compare our outcome, presence/absence of ear drainage, by our two independent variables, dornase alfa (Pulmozyme®) and Ofloxin

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Dornase Alfa (Pulmozyme®) | Ofloxin
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/22
Other Adverse Events (participants affected / at risk) | 11/19 | 11/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dornase Alfa (Pulmozyme®) (N=19) | Ofloxin (N=22)
Upper Respiratory Tract Infection/Viral Illness (Infections and infestations) | 5 | 4
Otitis Media (Ear and labyrinth disorders) | 2 | 5
Change in Hearing (Ear and labyrinth disorders) | 2 | 2
Cheek Laceration (Injury, poisoning and procedural complications) | 1 | 0
Allergies (Respiratory, thoracic and mediastinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No